CLINICAL TRIAL: NCT06680375
Title: A Phase 1/2, Randomized, Controlled Study to Evaluate the Reactogenicity, Safety, and Immunogenicity of an Investigational Flu Seasonal/SARS-CoV-2 Combination mRNA Vaccine in Adults
Brief Title: A Study of an Investigational Flu Seasonal/SARS-CoV-2 Combination Vaccine in Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 221542
Record Dates: First submitted 2024-11-06; First posted 2024-11-08 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: COVID-19
Keywords: Combination vaccine; Flu Seasonal; SARS-CoV-2 mRNA; Healthy younger adults; Healthy older adults; Safety; Reactogenicity; Immunogenicity; First time in humans
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This is an observer-blind study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- mRNA Flu/COVID-19 Dose 1 Group (Experimental): Participants receive one dose of investigational Flu mRNA vaccine composition in combination with a Dose 1 of a COVID-19 component and 1 dose of placebo on Day 1.
  Interventions: Combination Product: Flu Seasonal /SARS-CoV-2 mRNA Dose 1; Drug: Placebo
- mRNA Flu/COVID-19 Dose 2 Group (Experimental): Participants receive one dose of a Flu mRNA vaccine composition in combination with a Dose 2 of a COVID-19 component and 1 dose of placebo on Day 1.
  Interventions: Combination Product: Flu Seasonal /SARS-CoV-2 mRNA Dose 2; Drug: Placebo
- Flu+COVID-19 Group (Active Comparator): Participants receive one dose of a licensed Flu Seasonal vaccine and a licensed mRNA COVID-19 vaccine on Day 1.
  Interventions: Combination Product: Licensed Flu Seasonal; Combination Product: Licensed COVID-19 mRNA
- mRNA Flu Group (Active Comparator): Participants receive one dose of an investigational mRNA Flu Seasonal vaccine and 1 dose of placebo on Day 1.
  Interventions: Combination Product: Flu Seasonal mRNA; Drug: Placebo
- mRNA COVID-19 Dose 1 Group (Active Comparator): Participants receive one dose of Dose 1 investigational mRNA COVID-19 vaccine and 1 dose of placebo on Day 1.
  Interventions: Combination Product: SARS-CoV-2 mRNA Dose 1; Drug: Placebo
- mRNA COVID-19 Dose 2 Group (Active Comparator): Participants receive one Dose 2 investigational mRNA COVID-19 vaccine and 1 dose of placebo on Day 1.
  Interventions: Combination Product: SARS-CoV-2 mRNA Dose 2; Drug: Placebo

INTERVENTIONS:
Combination Product: Flu Seasonal /SARS-CoV-2 mRNA Dose 1 — A Flu mRNA vaccine composition in combination with Dose 1 of a COVID-19 component will be administered.
  Arms: mRNA Flu/COVID-19 Dose 1 Group
Combination Product: Flu Seasonal /SARS-CoV-2 mRNA Dose 2 — A Flu mRNA vaccine composition in combination with Dose 2 of a COVID-19 component will be administered.
  Arms: mRNA Flu/COVID-19 Dose 2 Group
Combination Product: Flu Seasonal mRNA — An investigational mRNA Flu Seasonal vaccine will be administered.
  Arms: mRNA Flu Group
Combination Product: SARS-CoV-2 mRNA Dose 1 — Dose 1 of an investigational mRNA COVID-19 vaccine will be administered.
  Arms: mRNA COVID-19 Dose 1 Group
Combination Product: SARS-CoV-2 mRNA Dose 2 — Dose 2 of an investigational mRNA COVID-19 vaccine will be administered.
  Arms: mRNA COVID-19 Dose 2 Group
Combination Product: Licensed Flu Seasonal — A licensed Flu Seasonal vaccine will be administered.
  Arms: Flu+COVID-19 Group
Combination Product: Licensed COVID-19 mRNA — A licensed mRNA COVID-19 vaccine will be administered.
  Arms: Flu+COVID-19 Group
Drug: Placebo — A placebo will be administered.
  Arms: mRNA COVID-19 Dose 1 Group; mRNA COVID-19 Dose 2 Group; mRNA Flu Group; mRNA Flu/COVID-19 Dose 1 Group; mRNA Flu/COVID-19 Dose 2 Group

SUMMARY:
This study will evaluate the reactogenicity, safety, and immune response of Flu Seasonal/SARS-CoV-2 mRNA (mRNA Flu/COVID-19) combination vaccine. The flu portion will target multiple strains of the flu virus, while the COVID-19 part will focus on the spike protein of the SARS-CoV-2 virus. Both parts of this vaccine have been tested individually before. This will be the first study to test the combined vaccine in humans in healthy adult participants.

DETAILED DESCRIPTION:
Click here to enter text.

ELIGIBILITY:
Inclusion Criteria:

* Participants, who, in the opinion of the investigator, can and will comply with the requirements of the protocol (e.g., completion of the eDiary, return for follow-up visits).
* Written informed consent obtained from the participant prior to performance of any study-specific procedure.
* A male or female 18-64 years of age (YA: 18-64) at the time of the study intervention administration.
* Participants must have a body mass index (BMI) >=18 kg/m² and less than equal to (<=) 40 kg/m2.
* Healthy participants or medically stable patients as established by medical history, clinical examination and (safety laboratory assessments). Participants with chronic medical conditions with or without specific treatment (e.g., chronic metabolic, cardiac, pulmonary, renal, hepatic, neurologic, and hematologic diseases) are allowed to participate in this study, if considered by the investigator as medically stable. A stable medical condition is defined as disease not requiring significant change in therapy or hospitalization for worsening disease during 3 months before enrolment.
* Prior receipt of a COVID-19 vaccine. This may be from a completed primary vaccination series or booster dose(s) of an approved or authorized COVID-19 vaccine. The last COVID-19 vaccination must have been received at least 90 days prior to randomization.
* Women of non-childbearing potential may be enrolled in the study.
* Women of childbearing potential may be enrolled in the study if the participant:

  * has practiced adequate contraception for 4 weeks prior to study intervention administration, and
  * has a negative pregnancy test on the day of study intervention administration, and has agreed to continue adequate contraception for at least 8 weeks after completion of the study intervention administration.

Exclusion Criteria:

Medical conditions

* Any clinically significant hematological, biochemical laboratory abnormality.
* Participant tested positive for influenza by local health authority-approved testing methods within 180 days prior to Day 1.
* A documented history of confirmed SARS-CoV-2 infection within 90 days before study vaccination.
* Has had known close contact with anyone who had confirmed influenza or a confirmed SARS-CoV-2 infection within 2 weeks before study vaccination.
* Current or past malignancy, unless completely resolved without clinically significant sequelae (e.g., no evidence of disease following successful treatment of basal cell carcinoma cases are allowed) for >5 years.
* Has any medical disease or psychiatric condition that, in the opinion of the investigator, precludes study participation because it would place the participant at an unacceptable risk of injury, would render them unable to meet the requirements of the protocol, or may interfere with successful completion of the study.
* Has a bleeding disorder (e.g., factor deficiency, coagulopathy, or platelet disorder), or prior history of significant bleeding or bruising following IM injections.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* Any history of an immunosuppressive or immunodeficient condition resulting from disease (e.g., HIV infection or congenital immunodeficiency).
* Has a history of hypersensitivity or severe allergic reaction including anaphylaxis, generalized urticaria, angioedema, and other significant reactions to any previous mRNA or non-mRNA vaccine or any component of the study intervention(s) (including polyethylene glycol, egg proteins and aminoglycoside antibiotics)
* History of uncontrolled neurological disorders or seizures, including Guillain-Barré syndrome (within 6 weeks of receiving any vaccine) and Bell's Palsy, with the exception of febrile seizures during childhood.
* History of or current suspicion of myocarditis or pericarditis (including following administration of an mRNA vaccine); or idiopathic cardiomyopathy, or presence of any medical condition that increases the risk of myocarditis or pericarditis, including cocaine abuse, cardiomyopathy, endomyocardial fibrosis, hypereosinophilic syndrome, hypersensitivity myocarditis, eosinophilic granulomatosis with polyangiitis and persistent myocardial infection.
* Any other clinical condition that, in the opinion of the investigator, might pose additional risk to the participant due to participation in the study.

Prior/Concomitant therapy

* Use of any investigational or non-registered product (drug, vaccine or invasive medical device) other than the study intervention(s) during the period beginning 28 days before the dose of study intervention(s) (Day -28 to Day 1), or their planned use during the study period.
* Administration of any mRNA-based vaccine in the period starting 28 days (Day -28) before study intervention administration.
* Administration of any influenza vaccine within 180 days before enrolment or planned administration within 28 days (Day 29) after the study intervention administration.

Administration of a vaccine not foreseen by the study protocol in the period starting 28 days (Day -28) before the study intervention administration or planned administration within 28 days (Day 29) after the study intervention administration.

* Chronic administration of immune-modifying drugs (defined as more than 14 consecutive days in total) and/or planned use of long-acting immune-modifying treatments at any time up to the end of the study.

  * Up to 3 months prior to the study intervention administration and up to the end of study: For corticosteroids, this will mean prednisone equivalent >=-20 mg/day. Inhaled, intra-articular and topical corticosteroids are allowed. If systemic corticosteroids have been administered short term (<14 days) for treatment of an acute illness, participants should not be enrolled into the study until corticosteroid therapy has been discontinued for at least 28 days before study vaccine administration.
  * Up to 3 months prior to study intervention administration and up to the end of the study: long-acting immune-modifying drugs including among others immunotherapy (e.g., TNF-inhibitors), monoclonal antibodies, antitumoral medication.
* Administration of immunoglobulins and/or any blood products or plasma derivatives within 3 months before study vaccination through end of study.

Prior/Concurrent clinical study experience

• Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational intervention.

Other exclusion criteria

* Participant is pregnant or has a positive pregnancy test result at Visit 1.
* Participant is breastfeeding or will (re)start breastfeeding between Day 1 (study vaccination) to 90 days after vaccination.
* Has a history of chronic alcohol consumption and/or drug abuse as deemed by the investigator to render the potential participant unable/unlikely to provide accurate safety reports or comply with study procedures.
* Participation of any study personnel or their immediate dependents, family, or household members.
* Participants with conditions precluding the assessment of local reactogenicity at the injection site (e.g, tattoos, scarring).
* Planned move during the study period that will prohibit participating in the study until study end.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 106 (Actual)
Dates: Start 2024-11-11 (Actual); Primary Completion 2025-06-09 (Actual); Study Completion 2025-06-09 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with increase in grading for at least one laboratory value from administration of study intervention | From Day 1 to Day 8
  Food and Drug Administration (FDA) toxicity grading scales for biochemistry hematology parameters are evaluated. Grades are defined as follows: Grade 1 - Mild; Grade 2 - Moderate; Grade 3 - Severe; Grade 4 -Potentially life threatening.
Percentage of participants with solicited administration site adverse events (AEs) | From Day 1 to Day 7
  The AEs considered are pain, redness, swelling and lymphadenopathy.
Percentage of participants with solicited systemic AEs | From Day 1 to Day 7
  The AEs considered are fever, headache, fatigue, myalgia, arthralgia and chills. Fever is defined as temperature greater than or equal to (>=) 38 °C/100.4°F regardless the location of measurement.
Percentage of participants with unsolicited AEs | From Day 1 to Day 28
  An unsolicited AE is an AE that was either not included in the list of solicited events or could be included in the list of solicited events but with an onset outside the specified period of follow-up for solicited events.
Percentage of participants with medically attended adverse events (MAAEs) | From Day 1 to Day 183 (study end)
  A MAAE is an AE for which the participant received medical attention including any symptom or illness requiring hospitalization, or an emergency room visit, or visit to/by a healthcare professional.
Percentage of participants with serious adverse events (SAEs) | From Day 1 to Day 183 (study end)
  A SAE is an AE which results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or other situations that are considered serious per medical or scientific judgment.
Percentage of participants with adverse events of special interest (AESIs) | From Day 1 to Day 183 (study end)
  The following events are considered as AESI in this study: severe hypersensitivity reactions within 24 hours after study intervention administration, myocarditis/pericarditis and potential immune-mediated diseases (pIMDs).
Geometric mean titer (GMT) ratio of antigen 1 antibody for investigational mRNA Flu/COVID-19 (pooled dose 1 and dose 2) and mRNA flu vaccines | At Day 29
GMT ratio of antigen 2 antibody for investigational mRNA Flu/COVID-19 (pooled dose 1 and dose 2) and mRNA flu seasonal vaccines | At Day 29
GMT ratio of serum neutralization titers against pseudovirus bearing spike from SARS-CoV-2 vaccine matched variant(s) for investigational mRNA Flu/COVID-19 (pooled dose 1 and dose 2) and mRNA COVID-19 vaccines | At Day 29

SECONDARY OUTCOMES:
GMT ratio of antigen 1 antibody for the investigational mRNA Flu/COVID-19 vaccines (dose 1 and 2) and Flu vaccines (pooled group) and licensed Flu vaccine co-administered with a licensed mRNA COVID-19 vaccine | At Day 29
GMT ratio of antigen 2 antibody for the investigational mRNA Flu/COVID-19 vaccines (dose 1 and 2) and Flu vaccines (pooled group) and licensed Flu vaccine co-administered with a licensed mRNA COVID-19 vaccine | At Day 29
GMT ratio of serum neutralization titers against pseudovirus bearing spike from SARS-CoV-2 vaccine matched variant(s) | At Day 29
  GMT ratio of serum neutralization titers against pseudovirus bearing spike from SARS-CoV-2 vaccine matched variant(s) will be evaluated for the investigational mRNA Flu/COVID-19 vaccines and COVID-19 with the same dose (pooled group) and licensed mRNA COVID-19 vaccine co-administered with a licensed Flu Seasonal vaccine.
GMTs of antigen 1 antibody for the investigational mRNA Flu/COVID-19 vaccines, mRNA Flu Seasonal vaccine and the licensed Flu Seasonal vaccine co-administered with a licensed mRNA COVID-19 vaccine | At Day 92 and Day 183 (Study end)
Geometric mean increase (GMI) in antigen 1 antibody for the investigational mRNA Flu/COVID-19 vaccines, mRNA Flu Seasonal vaccine and the licensed Flu Seasonal vaccine co-administered with a licensed mRNA COVID-19 vaccine | From Day 1 to Day 29, from Day 1 to Day 92 and from Day 1 to Day 183 (study end)
  GMI is defined as the geometric mean of the ratios of the post-vaccination titer over the Day 1 titer.
Seroconversion rate (SCR) of antigen 1 antibody for the investigational mRNA Flu/COVID-19 vaccines, mRNA Flu Seasonal vaccine and the licensed Flu Seasonal vaccine co-administered with a licensed mRNA COVID-19 vaccine | From Day 1 to Day 29, from Day 1 to Day 92 and from Day 1 to Day 183 (study end)
Seroprotection rate (SPR) of antigen 1 antibody for the investigational mRNA Flu/COVID-19 vaccines, mRNA Flu Seasonal vaccine and the licensed Flu Seasonal vaccine co-administered with a licensed mRNA COVID-19 vaccine | At Day 1, Day 29, Day 92, and Day 183 (study end)
GMTs of antigen 2 antibody for the investigational mRNA Flu/COVID-19 vaccines, mRNA Flu Seasonal vaccine and the licensed Flu Seasonal vaccine co-administered with a licensed mRNA COVID-19 vaccine | At Day 92 and Day 183 (study end)
GMI in antigen 2 antibody for the investigational mRNA Flu/COVID-19 vaccines, mRNA Flu Seasonal vaccine and the licensed Flu Seasonal vaccine co-administered with a licensed mRNA COVID-19 vaccine | From Day 1 to Day 29, from Day 1 to Day 92 and from Day 1 to Day 183 (study end)
  GMI is defined as the geometric mean of the ratios of the post-vaccination titer over the Day 1 titer.
SCR of antigen 2 antibody in for the investigational mRNA Flu/COVID-19 vaccines, mRNA Flu Seasonal vaccine and the licensed Flu Seasonal vaccine co-administered with a licensed mRNA COVID-19 vaccine | From Day 1 to Day 29, from Day 1 to Day 92 and from Day 1 to Day 183 (study end)
GMTs of serum neutralization titers against pseudovirus bearing spike from SARS-CoV-2 vaccine matched variant(s) | At Day 92, and Day 183 (study end)
  GMTs of serum neutralization titers against pseudovirus bearing spike from SARS-CoV-2 vaccine matched variant(s) will be evaluated for the investigational mRNA Flu/COVID-19 vaccines, mRNA COVID-19 vaccine and the licensed mRNA COVID-19 vaccine co-administered with a licensed Flu Seasonal vaccine
GMI of neutralization titers against pseudovirus bearing spike from SARS-CoV-2 vaccine matched variant(s) | At Day 29, Day 92, and Day 183 (study end)
  GMI is defined as the geometric mean of the ratios of the post-vaccination titer over the Day 1 titer. GMI of neutralization titers will be evaluated for the investigational mRNA Flu/COVID-19 vaccines, mRNA COVID-19 vaccine and the licensed mRNA COVID-19 vaccine co-administered with a licensed Flu Seasonal vaccine.
Percentage of participants with seroresponse of neutralization titers against pseudovirus bearing spike from SARS-CoV-2 vaccine matched variant(s) | At Day 29, Day 92, and Day 183 (study end)
  Seroresponse of neutralization titers against pseudovirus bearing spike from SARS-CoV-2 vaccine matched variant(s) will be evaluated for the investigational mRNA Flu/COVID-19 vaccines, mRNA COVID-19 vaccine and the licensed mRNA COVID-19 vaccine co-administered with a licensed Flu Seasonal vaccine.

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - GSK Investigational Site, Anniston, Alabama
  - GSK Investigational Site, Rolling Hills Estates, California
  - GSK Investigational Site, Hialeah, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Lenexa, Kansas
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Rochester, New York

IPD SHARING:
Plan to Share IPD: Yes
Study Sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or asset(s) with development terminated across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf